CLINICAL TRIAL: NCT01807910
Title: Phospholipid Endoplasmic Reticulum Stress in Nonalcoholic Fatty Liver Disease
Brief Title: ER Stress in NAFLD
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The study was not funded
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Charles R. Flynn, Assistant Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ER stress
Record Dates: First submitted 2013-03-05; First posted 2013-03-08 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Obesity; NAFLD
Keywords: Obesity; NAFLD; NASH; Steatosis
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fructose (Experimental): Participants will receive fructose (3g/kg/day) for 2 weeks.
  Interventions: Drug: methyl-D9-choline
- Glucose (Active Comparator): Participants will receive glucose (3g/kg/day) for 2 weeks.
  Interventions: Drug: methyl-D9-choline

INTERVENTIONS:
Drug: methyl-D9-choline — Subjects in both arms will be infused with methyl-D9-choline in order to assess the biosynthesis and kinetics of secretory lipoprotein phospholipids.

SUMMARY:
The investigators overall hypothesis is that exacerbation of endoplasmic reticulum (ER) stress in the liver is associated with significant alterations in phosphatidylcholines that drive the NASH phenotype in obese humans. The investigators plan to examine this hypothesis in a well-characterized cohort of obese subjects that are scheduled for bariatric surgery. Methyl-D9-choline chloride will be infused before and after a 2-week high fructose or glucose feeding to determine the biosynthesis and kinetics of secretory lipoprotein phospholipids. It is proposed that phospholipid metabolism play an important role in the pathogenesis or etiology of fatty liver in non-alcoholic conditions through mechanisms that invoke ER and oxidative stress responses.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory females age 30-60 years old
* Women of all ethnic groups
* BMI≥35 kg/m2
* Approval for Roux-en-Y gastric bypass or sleeve gastrectomy.

Exclusion Criteria:

* Smoking >7 cigarettes per day
* Previous malabsorptive or restrictive intestinal surgery
* Pregnant or breastfeeding
* Recent history of neoplasia (<5 years ago)
* Malabsorptive syndromes
* Inflammatory intestinal disease
* Patients with established organ dysfunction
* Diagnosis of type 1 or type 2 diabetes mellitus or current use of anti-diabetic medication (last 30 days; last 60days for thiazolidinediones)
* Diagnosed hyperbetalipoproteinemia or hypobetalipoproteinemia
* Patients on cholesterol lowering medicines
* Vegan diet
* Hepatic fat content <10% by MRI
* Inability to comply with study protocol such as unable to make study visits or be available daily for phone contact
* Any condition which would interfere with MRI or PET studies, e.g. claustrophobia, cochlear implant, chronic back pain limiting ability to lay flat, metal fragments in eyes, cardiac pacemaker, neural stimulator, tattoos with iron pigment and metallic body inclusions or other metal implanted in the body which may interfere with MRI scanning.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Net hepatic phospholipid production | Baseline and 2 weeks
  Net hepatic phospholipid production will be determined using [11C]choline dynamic Positron Emission Tomography (PET) before and after high fructose feeding for two weeks. A similar group of control obese subjects will undergo the same procedures before and after two weeks isocaloric glucose feeding.

SECONDARY OUTCOMES:
Kinetics of secretory lipoprotein phospholipids | Baseline and 2 weeks
  The biosynthesis and kinetics of secretory lipoprotein phospholipids will be determined using methyl-D9-choline chloride infusion before and after high fructose (or glucose) feeding.

OTHER OUTCOMES:
Changes in zonation of phospholipids and PEMT in liver tissues | 60 months
  Changes in zonation of phospholipids and PEMT in liver tissues acquired from the same subjects intraoperatively during bariatric surgery will be assessed using MALDI-IMS.

CONTACTS AND LOCATIONS:
Overall Officials: Charles R Flynn, PhD, Principal Investigator — Vanderbilt University Medical Center; Naji N Abumrad, MD, Study Chair — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States